CLINICAL TRIAL: NCT00296309
Title: A Multicentre, Randomised, Open Clinical Study to Compare the Efficacy and Safety of a Combination of Tacrolimus and Mycophenolate Mofetil Based Regimen With or Without Induction in Elderly Recipients Undergoing Kidney Transplantation
Brief Title: Comparing Efficacy & Safety of Tacrolimus & MMF With/Without Induction in the Elderly Following Kidney Transplantation.
Acronym: SENIOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FG-506-02-42
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Kidney Transplantation
Keywords: Tacrolimus; Kidney Transplantation; Immunosuppression; Adult; Treatment Outcomes
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Tacrolimus
- 2 (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Immunosuppression

SUMMARY:
Primary objective of this study is to compare the renal function as well as the incidence of renal dysfunction, the incidence of death, graft loss and acute rejection. Secondary Objective is to compare the efficacy and safety profiles of the two regimens in elderly renal transplanted patients.

DETAILED DESCRIPTION:
The use of tacrolimus-based primary immunosuppression in elderly renal transplant recipients is efficacious and safe, particularly in combination with MMF, and seems to be associated with lower mortality and graft loss rates than classic cyclosporin protocols. Nevertheless, the efficacy and safety of tacrolimus in monotherapy, double or triple therapy with MMF, as well as the induction therapy with the new anti-IL2 receptor antibodies have not been adequately used in controlled trials in the elderly renal transplant patient. There is only scarce information on age-associated immune responsiveness and only a few aged-adapted immunosuppressive regimens have been described.

ELIGIBILITY:
Inclusion Criteria:

* Patients with minimum 60 years of age and end stage kidney disease who are suitable candidates for primary renal transplantation or retransplantation are eligible for the study. Patients receiving a kidney transplant, from a cadaveric or living donor (not HLA identical) with compatible ABO blood type can be included.

Exclusion Criteria:

* Patient has an immunological high risk
* Cold ischemia time greater than 30 hours.
* Patient has significant liver disease
* Patient is allergic or intolerant to study medication
* Patient or donor is known to be HIV positive.
* Patient with malignancy or history of malignancy
* Patient has significant, uncontrolled concomitant infections

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2004-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Renal function measured by creatinine clearance | 6 months

SECONDARY OUTCOMES:
Acute rejection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Physician, Study Director — Astellas Pharma Europe B.V.
Locations (31):
- Belgium (2):
  - Brussels
  - Leuven
- France (10):
  - Bordeaux
  - Clermont-Ferrand
  - Créteil
  - Le Kremlin-Bicêtre
  - Montpellier
  - Nice
  - Suresnes
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (12):
  - Berlin
  - Cologne
  - Essen
  - Freiberg
  - Halle
  - Hanover
  - Jena
  - Leipzig
  - Lübeck
  - München
  - Münster
  - Rostock
- Utrecht, Netherlands
- Spain (2):
  - Madrid
  - Santander
- Zurich, Switzerland
- United Kingdom (3):
  - Belfast
  - Cambridge
  - Nottingham

REFERENCES:
- See also: Link to FDA Website — http://www.accessdata.fda.gov/scripts/cder/drugsatfda